CLINICAL TRIAL: NCT00340054
Title: Assessment of Occupational EMF Exposure - Validation of Interview Procedures Used in Brain Tumor Study
Brief Title: Developing Interview Questions to Estimate Workplace Exposure to Electric and Magnetic Fields
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: 99906013; 06-C-N013; 999906013; CDR0000551595; NCT00481910 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms

INTERVENTIONS:
Other: questionnaire administration
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Electric and magnetic fields may increase the risk of cancer. Developing interview questions that accurately estimate a person's exposure to electric and magnetic fields may help doctors learn about the long-term effects of workplace exposure.

PURPOSE: This clinical trial is developing interview questions that can be used in estimating workplace exposure to electric and magnetic fields.

DETAILED DESCRIPTION:
OBJECTIVES:

* Validate an interview-based electric and magnetic field exposure (EMF) assessment algorithm against measurements of the time-weighted average magnetic field magnitude used in previous epidemiologic studies.
* Calibrate the parameters in the algorithm in order to improve the exposure estimates.
* Correlate EMF exposure estimates from the algorithm with biologically based metrics measured by new instrumentation.

OUTLINE: Participants respond to questions during a 5- to 15-minute telephone interview concerning workplace exposure to electric and magnetic (EMF) fields. Data is collected during the interview using an exposure assessment algorithm designed to estimate EMF workplace exposure based on participants' responses. The interview-based estimates are then validated against actual field measurements of magnetic field exposure captured by Emdex multiwave monitors located at participating sites.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following occupation criteria:

  * Three occupations that primarily work in offices at Lawrence Livermore National Laboratories (LLNL)
  * Three occupations that do nonelectric manual work (e.g., machinists and laborers) at LLNL

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2005-10; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Validation of an interview-based electric and magnetic field (EMF) exposure assessment algorithm
Calibration of algorithm parameters
Correlation between EMF exposure estimates from the algorithm with biologically based metrics measured by new instrumentation

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Coble, DSc, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Exponent, Inc., Menlo Park, California
  - National Institute for Occupational Safety and Health, Cincinnati, Ohio

REFERENCES:
- [Background] Kelsh MA, Kheifets L, Smith R. The impact of work environment, utility, and sampling design on occupational magnetic field exposure summaries. AIHAJ. 2000 Mar-Apr;61(2):174-82. doi: 10.1080/15298660008984526. PMID 10782189